CLINICAL TRIAL: NCT04543149
Title: Evaluation of Immune Cells in Patients With Granulomatous Mastitis
Brief Title: Immune Cells in Patients With Granulomatous Mastitis
Status: Completed | Type: Observational
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ufuk Oguz Idiz, Assoc. Prof. MD, Istanbul Training and Research Hospital
Other Study IDs: Granulomatous mastitis cell
Record Dates: First submitted 2020-09-03; First posted 2020-09-09 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Granulomatous Mastitis
Keywords: Mastitis; immunophenotyping; Flow-cytometry
MeSH Terms: conditions — Granulomatous Mastitis; Mastitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Patients with idiopathic granulomatous mastitis
  Interventions: Diagnostic Test: Flow cytometric immunophenotyping
- Control: Healthy volunteers
  Interventions: Diagnostic Test: Flow cytometric immunophenotyping

INTERVENTIONS:
Diagnostic Test: Flow cytometric immunophenotyping — To evaluate T cell subsets and monocyte

SUMMARY:
Granulomatous mastitis is a rare, chronic, benign inflammatory disease of the breast that plays a role in many varying etiologies, including infectious and non-infectious causes. Etiological reasons were examined in various studies, but neither etiology nor definite criteria for diagnosis were found. Our aim in this study is to examine the role of immunophenotyping in differentiating the etiology of granulomatous mastitis and using it as a prognostic marker.

DETAILED DESCRIPTION:
Granulomatous mastitis is a rare, chronic, benign inflammatory disease of the breast that plays a role in many varying aetiology, including infectious and non-infectious causes. This disease can clinically and radiographically mimic breast cancer, which can pose a diagnostic challenge as well as concern during evaluation. A nonspecific inflammatory response, 'granuloma' is defined as necrosis or infiltration of other inflammatory leukocytes, with or without mononuclear phagocyte collection. It is thought to be caused by infectious agents or foreign substances that activate the immune system, leading to granuloma formation. Some of the known inflammatory etiologies of granulomatous mastitis are autoimmune diseases such as tuberculosis (most commonly caused by Mycobacterium tuberculosis), sarcoidosis, fungal infection and granulomatosis with polyangiitis and giant cell arteritis. These diseases cannot be distinguished clinically, pathologically, and radiographically from idiopathic granulomatous mastitis.In this study, we aimed to investigate lymphocyte subtypes in patients with granulomatous mastitis and to evaluate the differences in cell populations and its usability as a predictive marker in diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with granulomatous mastitis

Exclusion Criteria:

* Cancer Patients
* Patients with known immunodeficiency
* Pregnancy
* Patient diagnosed with tuberculosis

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Granulomatous mastitis is observed in female patients.
Study Population: In case group patients with granulomatous mastitis will be included to the study. During diagnasis if the patient is diagnosed with tuberculosis, she will be excluded from the study.
  Also healty volunteers who don't have breast lesions are control group.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-10 (Actual)

PRIMARY OUTCOMES:
To evaluate T cell subsets and monocyte ratio | 3 months
  CD3 (+) lymphocytes, CD4 (+) lymphocytes, CD 8 (+) lymphocytes, CD 3(-)/CD16 (+) NK cell ratio, CD14 (+) lymphocytes, and HLA-DR positivity on CD14 (+) cells

CONTACTS AND LOCATIONS:
Overall Officials: Ufuk Oguz Idiz, Assoc.Prof., Principal Investigator — Istanbul Training and Research Hospital
Locations (1):
- Istanbul Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barreto DS, Sedgwick EL, Nagi CS, Benveniste AP. Granulomatous mastitis: etiology, imaging, pathology, treatment, and clinical findings. Breast Cancer Res Treat. 2018 Oct;171(3):527-534. doi: 10.1007/s10549-018-4870-3. Epub 2018 Jul 3. PMID 29971624
- [Background] Skandarajah A, Marley L. Idiopathic granulomatous mastitis: a medical or surgical disease of the breast? ANZ J Surg. 2015 Dec;85(12):979-82. doi: 10.1111/ans.12929. Epub 2014 Nov 26. PMID 25424519